CLINICAL TRIAL: NCT03659149
Title: An Open-label, Randomized, Fasted, Single-dose, Three-way Crossover Study to Compare the Pharmacokinetics and Safety Between Administration of CKD-333 and Coadministration of CKD-330 and D086 in Healthy Male Adults
Brief Title: Pharmacokinetics and Safety Profile of CKD-333
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 170PK18015
Record Dates: First submitted 2018-09-03; First posted 2018-09-06 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-08

CONDITIONS: Hypertension; Dyslipidemias
Keywords: Hypertension; Dyslipidemias; CKD-333
MeSH Terms: conditions — Hypertension; Dyslipidemias | interventions — Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (Experimental): Period 1: Test drug 1(CKD-333 formulation I) Period 2: Test drug 2(CKD-333 formulation II) Period 3: Reference drug(CKD-330 + D086)
  Interventions: Drug: CKD-333 formulation I; Drug: CKD-333 formulation II; Drug: CKD-330+D086
- Group 2 (Experimental): Period 1: Test drug 1(CKD-333 formulation I) Period 2: Reference drug(CKD-330 + D086) Period 3: Test drug 2(CKD-333 formulation II)
  Interventions: Drug: CKD-333 formulation I; Drug: CKD-333 formulation II; Drug: CKD-330+D086
- Group 3 (Experimental): Period 1: Test drug 2(CKD-333 formulation II) Period 2: Reference drug(CKD-330 + D086) Period 3: Test drug 1(CKD-333 formulation I)
  Interventions: Drug: CKD-333 formulation I; Drug: CKD-333 formulation II; Drug: CKD-330+D086
- Group 4 (Experimental): Period 1: Test drug 2(CKD-333 formulation II) Period 2: Test drug 1(CKD-333 formulation I) Period 3: Reference drug(CKD-330 + D086)
  Interventions: Drug: CKD-333 formulation I; Drug: CKD-333 formulation II; Drug: CKD-330+D086
- Group 5 (Experimental): Period 1: Reference drug(CKD-330 + D086) Period 2: Test drug 1(CKD-333 formulation I) Period 3: Test drug 2(CKD-333 formulation II)
  Interventions: Drug: CKD-333 formulation I; Drug: CKD-333 formulation II; Drug: CKD-330+D086
- Group 6 (Experimental): Period 1: Reference drug(CKD-330 + D086) Period 2: Test durg 2(CKD-333 formulation II) Period 3: Test drug 1(CKD-333 formulation I)
  Interventions: Drug: CKD-333 formulation I; Drug: CKD-333 formulation II; Drug: CKD-330+D086

INTERVENTIONS:
Drug: CKD-333 formulation I — 1 tablet administered before the breakfast(single-dose)
  Other Names: Test drug
Drug: CKD-333 formulation II — 1 tablet administered before the breakfast(single-dose)
  Other Names: Test drug
Drug: CKD-330+D086 — 2 tablet administered before the breakfast(single-dose)
  Other Names: Reference drug

SUMMARY:
Compare the pharmacokinetic characteristics and safety between CKD-333 tablet and CKD-330, D086 combination

DETAILED DESCRIPTION:
An open-label, randomized, fasted, single-dose, three-way crossover study to compare the pharmacokinetic characteristics and safety between administration of CKD-333 and coadministration of CKD-330 and D086 in healthy male adults

ELIGIBILITY:
Inclusion Criteria:

1. Between 19 aged and 45 aged in healthy male adult
2. Body weight more than 50kg and within ideal body weight ±20%

Exclusion Criteria:

1. Have clinical significant medical history or disease that cardiovascular system, respiratory system, kidney, endocrine system, hematological system, digestive system , mental illness
2. Have a gastrointestinal disease history that can effect drug absorption or surgery
3. SBP(Systolic Blood pressure)≥140mmHg or SBP<90mmHg, DBP(Diastolic Blood Pressure(≥90mmHg or DBP<60mmHg

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-12 (Actual)

PRIMARY OUTCOMES:
AUCt(Area under the plasma drug concentration-time curve) PK of Candesartan, Amlodipine, Atorvastatin | 0~72hours
Cmax(Maximum plasma concentration of the drug in plasma) of Candesartan, Amlodipine, Atorvastatin | 0~72hours

SECONDARY OUTCOMES:
AUCinf(Area under the plasma concentration-time curve from time t to infinity) of Candesartan, Amlodipine, Atorvastatin, 2-hydroxy-atorvastatin | 0~72hours
Tmax(Time to reach the maximum concentration) of Candesartan, Amlodipine, Atorvastatin, 2-hydroxy-atorvastatin | 0~72hours
t1/2(Time for Cmax to drop in half) of Candesartan, Amlodipine, Atorvastatin, 2-hydroxy-atorvastatin | 0~72hours
CL/F(Apparent clearance) of Candesartan, Amlodipine, Atorvastatin, 2-hydroxy-atorvastatin | 0~72hours
Vd/F(Apparent volume of distribution) of Candesartan, Amlodipine, Atorvastatin, 2-hydroxy-atorvastatin | 0~72hours

CONTACTS AND LOCATIONS:
Overall Officials: Seunghun Han, Ph.D., Principal Investigator — Department of Clinical Pharmacology, Seoul ST.Mayr's Hospital
Locations (1):
- Seoul Saint Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No